CLINICAL TRIAL: NCT06667206
Title: Earlier Prime-BOOST Schedule to Improve MEasles Protection in High Burden Settings
Acronym: BoostMe
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: St George's, University of London (Other); MU-JHU CARE (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OVG2022/06
Record Dates: First submitted 2023-12-19; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2023-12

CONDITIONS: Measles
Keywords: measles-rubella vaccine
MeSH Terms: conditions — Measles

STUDY DESIGN:
Intervention Model Description: Equal numbers of participants are randomised to 3 arms.
Masking Description: All participants receive the same vaccines but are randomised to the timing of administration of the vaccines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: 6 and 12 months (Experimental): Early Prime-Boost schedule: Measles vaccines given at 6 and 12 months of age
  Interventions: Biological: Licenced Measles-Rubella vaccine
- Group B: 9 and 18 months (standard schedule) (Experimental): Standard schedule: Measles vaccines given at 9 and 18 months of age
  Interventions: Biological: Licenced Measles-Rubella vaccine
- Group C: 6 and 18 months (Experimental): Early Prime schedule: Measles vaccines given at 6 and 18 months of age
  Interventions: Biological: Licenced Measles-Rubella vaccine

INTERVENTIONS:
Biological: Licenced Measles-Rubella vaccine — Licenced Measles-Rubella vaccine provided by the Ugandan EPI programme

SUMMARY:
This is a phase IIb clinical trial investigating the non-inferiority of immune responses in children given two doses of measles vaccine at different timepoints. The study will randomise 450 children to 3 groups: group A will receive measles containing vaccine (MCV) at 6 and 12 months ; group B at 9 and 18 months; Group C at 6 and 18 months.

DETAILED DESCRIPTION:
Two doses of measles containing vaccine (MCV) are recommended in young children with the first dose given at different times depending on the setting. In low-incidence settings the MCV1 is given at 12 months of age or later as more infants over 12 months of age respond to MCV1 due to the absence of maternal antibody interference and an overall better immune response due to the maturation of the infant immune system. In high measles incidence settings MCV1 is given earlier at 9 months of age as there is no remaining protection from maternal antibody at this age and risk of infection if unvaccinated can be high. However, in children born with low levels or rapid decay of maternal antibody, the 9-month timing for MCV1 means the infant may be susceptible to infection for some months prior to vaccination. Therefore, in settings of high infant measles incidence, an early first dose at 6 months of age may bridge this susceptibility gap.

Our study will assess differences in protective levels of measles antibody in children randomised to receive early (6 months) or standard (9 months) MCV1 in a high incidence measles setting, and early (12 months) or standard (18 months) booster vaccines, in those who are given early MCV1. There will be 5 blood draws over 2 years. The study will compare children who received a) two doses of measles vaccine at 6 and 18 months with 9 and 18 months, and b) two doses of measles vaccine at 6 and 12 months compared with 6 and 18 months.

The study is funded by the Bill & Melinda Gates Foundation (INV-048650)

ELIGIBILITY:
1. Trial Participants Children aged 6 months (23 - 28 weeks) at time of screening
2. Inclusion Criteria

   * Aged 6 months (23 - 28 weeks) at time of screening
   * Received all previous vaccines as per country Expanded Programme of Immunization (EPI) schedule, verified by child health card
   * Parents/caretakers willing to give informed consent for their and their children's participation and stay in the geographical area where the study would be conducted
3. Exclusion Criteria

The participant may not enter the trial if any of the following apply:

* Child not healthy enough to be vaccinated in the opinion of the investigator
* Recent family history of measles infection (since birth)
* Previous receipt of any measles vaccination
* A family history of congenital or hereditary immunodeficiency other than HIV
* Receipt of more than 1 week of immunosuppressant or immune modifying drugs e.g. high dose steroids.
* Major congenital defects or serious chronic illness that in the opinion of the investigator are likely to modify immune responses or the ability to comply with the requirements of the study.
* History of any neurological disorders or seizures
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period
* Other abnormalities or medical history that contraindicated measles vaccination

Ages: 23 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Protective measles antibody concentrations at 2.5 years of age | 2.5 years of age
  Proportion of participants with protective levels of measles neutralising antibodies (PRNT>120mIUL)
Local and systemic reactions | 7 days post each vaccination
  Reactogenicity profile from diary cards
Serious Adverse Events | 2 years: (from baseline vaccination until 2 year follow up visit)

SECONDARY OUTCOMES:
Measles plaque reduction neutralisation titre (PRNT) and immunoglobulin G (IgG) concentration | one month after first dose
  Measles PRNT and IgG concentrations one month after first dose in infants receiving an early (6 months) compared to standard (9 month) dose of MCV
The effect of maternal human immunodeficiency virus (HIV) infection | one month after first dose and second dose
  Infant PRNT and IgG responses post MCV1 and MCV2 in children of mothers with and without HIV
The effect of maternal antibodies on infant immune response | pre-vaccination, 4 weeks after the first dose, 4 weeks after the second dose
  Relationship between baseline titres (pre vaccination) and 4 week post-vaccination titres for PRNT, Measles IgG, and measles ELISpot.
Immune response to rubella component of the vaccine | 4 weeks after a first and second dose
  Anti-rubella IgG

OTHER OUTCOMES:
Public perceptions of measles immunisation | Baseline until 2 year follow up visit
  Focus group interviews with the public and parents/guardians of enrolled children

CONTACTS AND LOCATIONS:
Locations (1):
- Makarere University - Johns Hopkins University Collaboration, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes